CLINICAL TRIAL: NCT03426189
Title: HIV Persistence in Lymph Node Tissue and Peripheral Blood: The Role of Immune Checkpoints
Brief Title: HIV Persistence in Lymph Node and Peripheral Blood
Acronym: HIV-PRADA
Status: Completed | Type: Observational
Sponsor: University of Melbourne (Other)
Collaborators: amfAR, The Foundation for AIDS Research (Other); University of California, San Francisco (Other); Monash University (Other); Université de Montréal (Other); The Avenue Hospital (Unknown); Oregon Health and Science University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Sharon Lewin, Director, The Peter Doherty Institute for Infection and Immunity, University of Melbourne
Other Study IDs: 1646930
Record Dates: First submitted 2017-12-03; First posted 2018-02-08 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: HIV-1-infection
Keywords: HIV; Latent reservoir; Leukapheresis; Inguinal lymph node biopsy; Immune checkpoint; PD1; CTLA4
MeSH Terms: interventions — Leukapheresis; Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Blood (CD4+ T cells, CD8+ T cells; plasma)
  * Lymph node biopsy (CD4+ T cells, CD8+ T cells)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV infected individuals on long term ART: * Leukapheresis
  * Lymph node biopsy
  Interventions: Procedure: Leukapheresis; Procedure: Lymph node biopsy

INTERVENTIONS:
Procedure: Leukapheresis — Blood will be taken by a needle inserted into a vein in one arm and processed through a machine, which spins the blood so that the white blood cells will be separated out of the machine for purposes of this research. The rest of the blood will be returned through a needle in the other arm.
Procedure: Lymph node biopsy — Ultrasound will be used to localize the position of one lymph node in the groin. Under a light general anesthetic, one lymph node will be removed.

SUMMARY:
The aim of this project is to determine whether latent HIV is enriched in cells expressing certain proteins (receptors) on their surface and whether it is possible to eliminate these cells through the use of drugs that specifically target these proteins. Lymph nodes are known to contain very high numbers of HIV infected cells.

DETAILED DESCRIPTION:
Combination antiretroviral therapy (ART) has significantly improved the immune function of HIV infected individuals and has transformed a fatal disease into a chronic infection for those with access to ART. Despite suppressing HIV-1 replication, ART is not curative and nearly all HIV infected individuals experience viral rebound within weeks or months of discontinuing ART. This rebound is because HIV is able to hide in long-lived and proliferating CD4+ T cells, a specific type of cell, found in the immune system. The ability to hide is referred to as HIV latency.

One strategy towards eliminating the reservoir of latently infected cells is characterized by the use of latency reversing agents (LRA) to reverse HIV-1 latency. This exposes virus-expressing cells to the immune system and ART virus-mediated cell lysis or immune-mediated killing. Emerging data suggests that HIV-1 is enriched in cells expressing certain proteins known as immune checkpoints (IC). Immune checkpoint proteins play an important role in the regulation of the immune system. By blocking the immune checkpoint with drugs, this approach would allow the immune system to recognize HIV infected cells as foreign and thereby attack and kill the cell. Currently, there are licensed antibodies to the specific IC known as PD-1 (Programmed cell death protein 1) and CTLA4 (Cytotoxic T-Lymphocyte Associated Protein 4). These antibodies are in clinical use for the treatment of a range of malignancies.

Most of what is known about HIV-1 latency, reservoir composition, activation of HIV-1 by LRAs and viral enrichment in cells expressing IC in individuals on suppressive ART, is based on studies of peripheral blood T cells rather than lymphoid tissue. However, only 10% of the body's total CD4+T cell population is circulating at any one time. The rest of the CD4+ T cell population resides in the lymph nodes. In addition, cells that express IC are usually located in lymph nodes.

Using CD4+ T-cells from blood and lymph node tissue collected from HIV-infected individuals on ART, this study will examine if HIV is located in cell populations that express ICs and if blocking IC pathways can boost immune recognition of HIV infected cells.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Willing to undergo leukapheresis and lymph node biopsy
* Documented HIV-1 infection (antibody positive or detectable plasma HIV-1 RNA)
* Receiving combination ART
* HIV RNA < 50 copies/mL for > 3 years (Episodes of a single HIV plasma RNA 50-500 copies/mL will not exclude participation if the subsequent HIV plasma RNA was <50 copies/mL)

Exclusion Criteria:

* Unwillingness to follow protocol requirements
* Contraindications to LN biopsy or leukapheresis
* Current skin infection of inguinal area
* Known current lower extremity, gastrointestinal or genitourinary infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected individuals on long term antiretroviral therapy
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

PRIMARY OUTCOMES:
Frequency of HIV-1 in cells expressing CTLA4 and PD-1 in lymph node derived cells | Baseline only

SECONDARY OUTCOMES:
Frequency of HIV-1 in cells expressing CTLA4 and PD-1 in blood derived cells | Baseline only
Change in interferon gamma production in HIV specific T-cells following ex vivo blockade of PD-1 and CTLA4 | Baseline only
  Using blood and tissue from HIV infected individuals on ART, intracellular cytokine staining will be performed to detect interferon and other cytokines following stimulation with HIV pooled peptides

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Lewin, Principal Investigator — The Peter Doherty Institute for Infection and Immunity, University of Melbourne
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided